CLINICAL TRIAL: NCT06036979
Title: A Comparative Study Between Preoperative Erector Spinae Plane Block Versus Preoperative Paravertebral Plane Block in Decreasing Post Mastectomy Pain Syndrome. A Randomized Controlled Study.
Brief Title: Preoperative Erector Spinae Plane Block Versus Paravertebral Plane Block in Decreasing Post Mastectomy Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AP2303-301-0007
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Chronic Postoperative Pain
Keywords: PVPB, ESPB, prevention of PMPS
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Analgesics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Paravertebral Block Group (Active Comparator): This group will receive combined general anaesthesia with preoperative ultrasound guide paravertebral plane block
  Interventions: Procedure: Paravertebral plane block
- Erector Spinae Block Group (Active Comparator): This group will receive combined general anaesthesia with preoperative ultrasound guided erector spinae plane block
  Interventions: Procedure: Erector spinae plane block
- Control Group (Other): This group will receive balanced general anesthesia using intravenous (0.1mg/kg) morphine, 30 mg ketorlac and 1 gm paracetamol).
  Interventions: Drug: Intravenous morphine, ketorlac and paracetamol

INTERVENTIONS:
Procedure: Paravertebral plane block — With the patients are placed in the sitting position, counting down from C7 spinous process, a high frequency linear ultrasound probe is placed on the spinous process in the parasagittal plane at T5 level and then is slided laterally 2-3 cm to make the transverse processes clearly visualized . Under aseptic conditions, a 22-gauge block needle (50mm, B.Braun, Germany) is inserted using in-plane technique toward the paravertebral space, immediately above the pleura and below the superior costotransverse ligament. The position of the needle is confirmed by the descent of the pleura when injecting 2 to 3 ml of saline solution for hydrolocalization. Then 0.3ml/kg of bupivacaine 0.25% is injected under ultrasound guidance. Block success is defined as reduced sensitivity to cold and pinprick stimuli as compared with the contralateral side 20 minutes after local anesthetic injection.
  Other Names: PVPB
  Arms: Paravertebral Block Group
Procedure: Erector spinae plane block — With the patients are placed in the sitting position, counting down from C7 spinous process, a high frequency linear ultrasound probe is placed on the spinous process in the parasagittal plane at T5 level and then is slided laterally 2-3 cm to make the tips of the transverse processes clearly visualized . The following muscles seen from superficial to deep layer are trapezius, rhomboid major and erector spinae muscles. Under aseptic conditions, a 22-gauge block needle (50mm, B.Braun, Germany) is inserted using in-plane technique to reach the interfascial plane between the transverse process and the erector spinae muscle. Following confirmation of the accurate position of the needle tip with 3-5 ml normal saline solution, 0.3ml/kg of bupivacaine 0.25% is injected under ultrasound guidance. Block success is defined as reduced sensitivity to cold and pinprick stimuli as compared with the contralateral side 20 minutes after local anesthetic injection.
  Other Names: ESPB
  Arms: Erector Spinae Block Group
Drug: Intravenous morphine, ketorlac and paracetamol — • In the control group only we add 10mg intravenous morphine, 30 mg intravenous ketorlac and 1 gm intravenous paracetamol for analgesia.
  Other Names: IV analgesics
  Arms: Control Group

SUMMARY:
Breast cancer is considered the commonest malignancy affecting women with an incidence exceeding one million cases per year. Although it has a favorable prognosis with improved lines of treatment, some complications may still disturb the patient's life quality. One of these complications is post-mastectomy pain syndrome (PMPS) .Regional Anaesthesia (RA) is considered one of the most effective methods in reducing acute pain after breast surgeries, these include pectoral nerves block (PECS), serratus anterior plane block (SAPB), paravertebral plane block (PVPB) and erector spinae plane block (ESPB) . Our study is aiming for comparing the effect of preoperative PVPB versus preoperative ESPB in the prevention of PMPS in patients undergoing unilateral breast surgeries.

DETAILED DESCRIPTION:
Breast cancer is considered the commonest malignancy affecting women with an incidence exceeding one million cases per year. Although it has a favorable prognosis with improved lines of treatment, some complications may still disturb the patient's life quality. One of these complications is post-mastectomy pain syndrome (PMPS) ¹.

The International Association for Study of Pain (IASP) defines PMPS as chronic pain that persists more than 3 months in the anterior thorax, axilla &/or upper arm ². It is usually neuropathic in nature includes altered sensations such as dysesthesia, hypo or hyperesthesia, allodynia or particular qualities of dysesthesia e.g burning, dull aching sensations. It is usually of at least moderate intensity and may be either continuous or intermittent pain ³.

The etiology and mechanism of PMPS remain incompletely clear yet. Some risk factors are believed to be associated with PMPS, including the presence and intensity of postoperative pain, the type of surgery, younger women, prior history of other types of pain and adjuvant therapies like chemo or radiotherapy ⁴.

Regional Anaesthesia (RA) is considered one of the most effective methods in reducing acute pain after breast surgeries, these include pectoral nerves block (PECS), serratus anterior plane block (SAPB), paravertebral plane block (PVPB) and erector spinae plane block (ESPB) ⁵. Theoretically RA can minimize the development of PMPS by decreasing the afferent nociceptive input and central sensitization during the perioperative period, However clinically the role of RA in preventing PMPS is still under investigations ⁶.

PVPB includes injecting local anesthetic in the paravertebral space where the spinal nerves exit from the intervertebral foraminae. Paravertebral space is bounded by the parietal pleura, superior costotransverse ligament, vertebrae, intervertebral foraminae and the heads of the ribs ⁷. While ESPB includes injection of the local anesthetic in the fascial plane between the vertebral transverse processes and the erector spinae muscle ⁸.

Many studies were done in order to evaluate the efficacy of either ESPB or PVB in controlling acute postoperative pain after breast surgeries, some studies compared between them in controlling acute postoperative pain after breast surgeries ⁹. Also there are some studies that evaluate the effect of either ESPB or PVPB in the prevention of PMPS after breast surgeries ¹⁰, but still the comparison between the effect of preoperative ESPB versus the effect of preoperative PVPB in the prevention of PMPS in patients undergoing breast surgeries is still under investigated.

Our study is aiming for comparing the effect of preoperative PVPB versus preoperative ESPB in the prevention of PMPS in patients undergoing unilateral breast surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 60 years old.
* Female patients ASA ΙΙ, ΙΙΙ.
* Female patients scheduled for unilateral breast surgeries.

Exclusion Criteria:

* Patient refusal.
* Patients have sepsis
* Patients known to have allergy against local anesthetics.
* Patients with prior surgery in areas above or below the clavicle or in the axillary region.
* Patients with opioid dependence, alcohol or drug abuse.
* Patient with coagulopathy.
* Patients with psychiatric illness that prevent them from proper pain perception and assessment.
* ASA 4 or higher.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients ASA ΙΙ, ΙΙΙ between 18 and 60 years undergoing unilateral breast surgeries.
Enrollment: 51 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to assess the incidence of PMPS 3 months after surgery. | 3 months
  * A junior pain physician is blinded to all treatment groups and asks about symptoms of PMPS including (pain, tingling, numbness, shooting pain, pricking pain or unbearable itching), site (chest wall, armpit, arm, shoulder or surgical scar) and grading scale using the brief pain inventory (BPI).
  * Chronic pain is defined by a score of ≥ 3 on the single item (average pain) of the BPI.
  * The BPI consists of three domains: (1) Pain intensity measured using the visual analogue scale (VAS) of 0 (no pain) to 10 (worst pain). (2) Pain that interferes with daily activities measured using a scale of 0 (no interference) to 10 (complete restriction to daily activities). (3) Percentage of relief provided by pain treatments measured using a scale of 0 (complete relief) to 10 (no relief) by the NRS.

SECONDARY OUTCOMES:
• The prevalence of PMPS at 6 months. | 6 months
  • The prevalence of PMPS at 6 months.
• Assessment of acute postoperative pain. | 48 hours
  • Assessment of acute postoperative pain using VAS (0 for no pain, 10 for the worst pain) at 0, 4, 8, 24 and 48 hours postoperatively.
• Time to first needed morphine dose postoperatively, total 24-48 hours morphine consumption. | 48 hours .
  • Time to first needed morphine dose postoperatively, total 24-48 hours morphine consumption.
• PVPB and ESPB related complications. | 24 hours
  • PVPB and ESPB related complications (bupivacaine toxicity, pneumothorax).

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Ahmed, MS degree, Principal Investigator — National Cancer Institute, Egypt
Locations (1):
- NCIEGYPT, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be shared
Supporting Information: Study Protocol
Time Frame: 20 years
Access Criteria: Clinical trials.gov
URL: http://clinicaltrials.gov

REFERENCES:
- [Background] Harkouk H, Fletcher D, Martinez V. Paravertebral block for the prevention of chronic postsurgical pain after breast cancer surgery. Reg Anesth Pain Med. 2021 Mar;46(3):251-257. doi: 10.1136/rapm-2020-102040. Epub 2021 Jan 7. PMID 33414157
- [Background] Yuksel SS, Chappell AG, Jackson BT, Wescott AB, Ellis MF. "Post Mastectomy Pain Syndrome: A Systematic Review of Prevention Modalities". JPRAS Open. 2021 Oct 30;31:32-49. doi: 10.1016/j.jpra.2021.10.009. eCollection 2022 Mar. PMID 34926777
- [Background] Waltho D, Rockwell G. Post-breast surgery pain syndrome: establishing a consensus for the definition of post-mastectomy pain syndrome to provide a standardized clinical and research approach - a review of the literature and discussion. Can J Surg. 2016 Sep;59(5):342-50. doi: 10.1503/cjs.000716. PMID 27668333
- [Background] Gong Y, Tan Q, Qin Q, Wei C. Prevalence of postmastectomy pain syndrome and associated risk factors: A large single-institution cohort study. Medicine (Baltimore). 2020 May;99(20):e19834. doi: 10.1097/MD.0000000000019834. PMID 32443289
- [Background] Xin L, Hou N, Zhang Z, Feng Y. The Effect of Preoperative Ultrasound-Guided Erector Spinae Plane Block on Chronic Postsurgical Pain After Breast Cancer Surgery: A Propensity Score-Matched Cohort Study. Pain Ther. 2022 Mar;11(1):93-106. doi: 10.1007/s40122-021-00339-9. Epub 2021 Nov 26. PMID 34826113
- [Background] Zinboonyahgoon N, Patton ME, Chen YK, Edwards RR, Schreiber KL. Persistent Post-Mastectomy Pain: The Impact of Regional Anesthesia Among Patients with High vs Low Baseline Catastrophizing. Pain Med. 2021 Aug 6;22(8):1767-1775. doi: 10.1093/pm/pnab039. PMID 33560352
- [Background] Batra RK, Krishnan K, Agarwal A. Paravertebral block. J Anaesthesiol Clin Pharmacol. 2011 Jan;27(1):5-11. No abstract available. PMID 21804697
- [Background] Bonvicini D, Boscolo-Berto R, De Cassai A, Negrello M, Macchi V, Tiberio I, Boscolo A, De Caro R, Porzionato A. Anatomical basis of erector spinae plane block: a dissection and histotopographic pilot study. J Anesth. 2021 Feb;35(1):102-111. doi: 10.1007/s00540-020-02881-w. Epub 2020 Dec 19. PMID 33340344
- [Background] El Ghamry MR, Amer AF. Role of erector spinae plane block versus paravertebral block in pain control after modified radical mastectomy. A prospective randomised trial. Indian J Anaesth. 2019 Dec;63(12):1008-1014. doi: 10.4103/ija.IJA_310_19. Epub 2019 Dec 11. PMID 31879425
- See also: Comparative study between ultrasound guided erector spinae plane block versus paravertebral block for postoperative pain relief in patients undergoing unilateral modified radical mastectomy.AIMJ.2022. — https://aimj.journals.ekb.eg/article_230793.html